CLINICAL TRIAL: NCT00718055
Title: MR Skanning Med Leverspecifikt Oralt Kontraststof Sammenlignet Med CT Skanning Hos Colorectalcancer Patienter Med Levermetastaser
Brief Title: Magnetic Resonance Imaging (MRI) Using Liverspecific Oral Contrast Agent in Metastatic Colorectal Cancer Patients
Status: Withdrawn | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Vibeke Løgager, Herlev Hospital
Other Study IDs: KA-20060096
Record Dates: First submitted 2006-10-04; First posted 2008-07-18 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Neoplasm Metastasis; Liver; Colorectal Neoplasms; Magnetic Resonance Imaging; Contrast Media
Keywords: MRI; liverspecific; contrast; colorectal; metastases
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine whether MRI with manganese containing contrast agent detects more livermetastasis compared to CT scan

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved liver metastasis

Exclusion Criteria:

* pacemaker, metal in the body, claustrophobia, pregnancy, age below 18 years, psychiatry patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consekutive group of liver metastatic patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Løgager, M.D., Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen Uni. Hospital at Herlev dept. of Radiology, Herlev, Denmark